CLINICAL TRIAL: NCT02127606
Title: The Effect of Whole Body Vibration on Spasticity in Spinal Cord Injury Patients
Brief Title: The Effect of Whole Body Vibration on Spasticity in Persons With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-811-14
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Injury; Spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibration with tilt-table standing (Experimental): Participants in this arm will undergo alternating side-to-side, whole body vibration while standing on a tilt table for multiple treatments for a total of approximately 14 minutes for 3 sessions over 3 different days
  Interventions: Device: Vibration with tilt-table standing

INTERVENTIONS:
Device: Vibration with tilt-table standing
  Other Names: Galileo Tilt-Table; Galileo System; Vibrating platform; Whole-body vibration with tilt-table standing

SUMMARY:
Extended periods of tilt table standing have been observed to improve spasticity in individuals with spinal cord injury (SCI). The purpose of this study is to determine the effect of three sessions of whole body vibration while tilt table standing on spasticity in individuals with a complete or incomplete SCI above the neurological level of T10. Participants in this study will undergo whole body vibration while standing on a tilt table for a total of approximately 14 minutes for a total of 3 sessions on 3 separate days. Spasticity monitoring will be evaluated prior to and after the intervention with the Modified Penn Spasm Frequency Scale, an interview to obtain the individual's perception and impression of the effect of whole body vibration on the performance of activities of daily living, quality of life, pain scale, and global impression of change.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, 18 to 70 years of age, inclusive.
* The subject has neurological impairment secondary to a spinal cord injury that occurred at least six (6) months prior to the study that can be categorized as either a complete or incomplete spinal cord injury.
* The neurological level of lesion is above T10.
* The subject has self-reported stable moderate to severe spasticity (Modified Ashworth Score scale at or greater than a 2 at the hips or knees). Patients can be enrolled if on a stable dose of oral medications or intrathecal medications.
* The subject has self reported spasticity that negatively impacts his or her quality of life, impairs ability to perform activities of daily living (such as transfers, sitting, sleep, wheelchair use, and hobbies).
* The subject is able to stand with the assistance of a tilt table at a minimum of 70 degrees for 45 minutes without significant orthostasis or other adverse events or symptoms.
* The subject is able and willing to comply with the protocol.
* The subject is able to and has voluntarily given informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* The subject does not self report lower limb spasticity.
* The subject does not have self reported spasticity that negatively impacts his or her quality of life, impairs ability to perform activities of daily living (such as transfers, sitting, sleep, wheelchair use, and hobbies).
* The subject experiences symptoms consistent with infection, including but not limited to fever, chills, dysuria, gallbladder or kidney stones.
* The subject experiences pain that is not well controlled with consistent pain medication use.
* The subject has recent thromboembolism, diabetes mellitus, intractable hypertension or cardiac/pulmonary instability, internal fixation implants, acute thrombosis, pregnancy, acute inflammation of the locomotor system including active arthrosis or arthropathy, acute tendinopathy, acute hernia, acute discopathy, recent post-surgical wounds, epilepsy, rheumatoid arthritis, or recent fractures<6 months.
* The subject has a lumbar spinal hardware or artificial joints in the lower extremities.
* The subject is participating in any experimental studies that could alter the patient's spasticity.
* The subject has a concomitant brain injury or other cognitive deficits that would preclude following instructions.
* The subject has skin breakdown in areas receiving direct pressure during tilt table standing.
* The subject has any medical condition, including psychiatric disease that would interfere with the interpretation of the study results or the conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET) score after the third treatment | Participants will be followed for the duration of the 3 treatments, an expected average of 1 week

SECONDARY OUTCOMES:
Change from Baseline in the Pain Severity Numerical Rating Scale (NRS) score after the third treatment | Participants will be followed for the duration of the 3 treatments, an expected average of 1 week
Change from Baseline in the Penn Spasm Frequency Scale score after the third treatment | Participants will be followed for the duration of the 3 treatments, an expected average of 1 week

OTHER OUTCOMES:
Subject Global Impression of Change (SGIC) | After the third treatment, an expected average of 1 week
Adverse Events | Participants will be followed for the duration of the 3 treatments, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation; Trevor A. Dyson-Hudson, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States